CLINICAL TRIAL: NCT06224270
Title: Immunogenicity and Safety of the Adjuvanted Recombinant Zoster Vaccine in Adults with Inflammatory Bowel Disease on Biologic Immunosuppressive Therapies
Brief Title: Study of Response to Zoster Vaccine in Adults with Inflammatory Bowel Disease Treated with Medications
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1727; A534250 (Other: UW Madison); Protocol Version 6/14/2024 (Other: UW Madison)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases; IBD
Keywords: immunosuppressed; Recombinant Zoster Vaccine
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This is an open label, multicenter trial evaluating the safety and immunogenicity of recombinant herpes zoster vaccine in adults with IBD on immunosuppressive therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Adults with IBD (Experimental)
  Interventions: Biological: Adjuvanted Recombinant Zoster Vaccine (RZV)

INTERVENTIONS:
Biological: Adjuvanted Recombinant Zoster Vaccine (RZV) — The RZV vaccine is indicated for prevention of herpes zoster (HZ) in adults aged 18 years and older who are or will be at increased risk of HZ. Patients with IBD on immunosuppressive therapy are at increased risk for HZ.

SUMMARY:
This multi-center study will evaluate the safety and immune response to recombinant zoster vaccine (RZV) series in 264 patients with inflammatory bowel disease (IBD) on immunosuppressive therapy recruited from 6 study sites who can expect to be on study for up to 14 months.

DETAILED DESCRIPTION:
Study Visits:

* Visit 1 (V1) - day 1 - blood draw, RZV dose 1

  * Follow up (FU) 1 - between days 7-15
  * FU 2 - between days 22-29
* Visit 2 (V2) - between days 30-90 - RZV dose 2

  * FU 3 - V2 + 7-14 days
* Visit 3 (V3) - V2 + 21-50 days - blood draw
* Visit 4 (V4) - V2 + approximately 360 days - blood draw

Primary Objective:

• To demonstrate a 10% higher humoral immunogenicity following two doses of RZV in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.

Secondary Objectives:

* To evaluate the vaccine response rate (VRR) for anti-glycoprotein E (gE) humoral immune responses in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
* To characterize the anti-gE humoral immunogenicity at visit 1 (V1), visit 3 (V3), and visit 4 (V4) in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
* To evaluate the safety and reactogenicity following administration of RZV, up to 30 days post-last vaccination and during the entire post-vaccination follow-up period.
* To evaluate IBD activity following administration of RZV, up to 30 days post-last vaccination and during the entire post-vaccination follow-up period.

Tertiary/Exploratory Objectives:

* To characterize gE-specific CD4+ T-cell mediated immune responses in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
* To characterize gE-specific CD4+ T-cell mediated immune responses in patients on JAKs.
* To evaluate the VRR for anti-gE humoral immune responses in patients on Janus Kinase inhibitors (JAKs).
* To characterize the anti-gE humoral immunogenicity at V1, V3, and V4 in patients on JAKs.
* To determine the relationship between gut microbiota and response to RZV series.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between the ages of 19 and 85 years with a diagnosis of IBD based on standard clinical and histological criteria.
* Can provide appropriate written informed consent.
* Patient has a history of ulcerative colitis or Crohn's disease diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria.
* Patient is receiving one of the following treatments for their IBD:

  * Anti-TNF therapy (infliximab, adalimumab, certolizumab, or golimumab)

    * On anti-TNF monotherapy
    * Or anti-TNF therapy in combination with either 10mg of methotrexate or azathioprine at least 1.0mg/kg or 6-Mercaptopurine (6MP) 0.5mg/kg
  * Non-TNF therapy

    * On ustekinumab monotherapy or in combination with either 10mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
    * On vedolizumab monotherapy or in combination with either 10mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
    * On Risankizumab monotherapy or in combination with either 10mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
    * On mirikizumab monotherapy or in combination with either 10mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
  * Janus Kinase Inhibitor

    * On tofacitinib at least 5mg PO twice per day (BID)
    * On upadactinib at least 15mg PO BID
* Patient has been on stable biologic or JAK treatment for IBD for at least two months.
* Patient is in stable clinical remission

  o No recent corticosteroid prescription within the past two months.
* Female participant of non-childbearing potential (pre-menarche, current tubal ligation, hysterectomy, oophorectomy or post-menopause) and childbearing potential (if they had: practiced adequate contraception (include IUD or equivalent, hormonal contraceptive (e.g. pill, patch, ring, implant or an injection used consistently and that has reached full effect prior to the first dose of vaccine), hysterectomy and/or a bilateral tubal ligation or bilateral oophorectomy) for 1 month prior to vaccination and agrees to continue adequate contraception during the primary treatment period, and for 2 months after completion of the vaccination series). Non-pregnant females with a negative pregnancy test who are willing to practice adequate contraception during the primary treatment period, and for 2 months after completion of the vaccination series).

Exclusion Criteria:

* Patient cannot or will not provide written informed consent.
* Patient has been taking any dose of oral or intravenous steroids for more than 3 days within 2 months prior to immunization.
* Any confirmed or suspected HIV, primary immunodeficiency disease, disseminated or untreated malignancy, or systemic infection.
* Previous vaccination against HZ or varicella within the 12M preceding the first dose of RZV.
* Occurrence of varicella or HZ per clinical history, within the 12M preceding the first dose of RZV.
* Evidence or high suspicion, in the opinion of the investigator, of noncompliance or nonadherence to the use of induction and/or maintenance immunosuppressive therapies.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or study material and equipment.
* Any condition which, in the judgment of the investigator, would make intramuscular injection unsafe.
* Any condition which, in the judgment of the investigator, would make intramuscular injection unsafe.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) before Month 3 (i.e. 2 months after last dose of study V2).

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Concentrations of Anti-gE Antibodies | Visit 3 (between 50 and 140 days on study)
  Anti-gE antibody concentrations expressed as geometric mean concentrations (GMCs) at V3, following 2 doses of RZV, in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.

SECONDARY OUTCOMES:
Vaccine response rate (VRR) | Visit 3 (between 50 and 140 days on study)
  Vaccine response rate (VRR) with exact 95% confidence intervals at V3 in those on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
Seropositivity rate | Visit 1 (day 1), Visit 3 (between 50 and 140 days on study), Visit 4 (approximately 360 days)
  Seropositivity rate with exact 95% confidence interval (CI) at V1, V3, and V4 in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
Geometric Mean Concentrations of Anti-gE Antibodies | Visit 1 (day 1), Visit 3 (between 50 and 140 days on study), Visit 4 (approximately 360 days)
  Anti-gE antibody concentrations expressed as GMC with 95% CI at V1, V3, and V4 in patients on non-TNF biologic therapy compared to those on anti-TNF biologic therapy.
Number of Participants with Solicited Adverse Events (AEs) | Up to 7 days after Visit 1, up to 7 days after Visit 2
  Number and percentage of patients reporting each solicited local AE and each solicited systemic AE within 7 days (Days 1-7) after each dose and overall for all study groups.
  Solicited local AEs are: injection site pain, redness, swelling.
  Solicited systemic AEs are: fatigue, myalgia, arthralgia, headache, shivering/chills, fever and gastrointestinal symptoms (nausea, vomiting, diarrhea, abdominal pain).
Number of Participants with Unsolicited Adverse Events | up to 30 days after Visit 1, up to 30 days after Visit 2
  Number and percentage of patients reporting unsolicited AEs within 30 days (Days 1-30) after each dose and overall, for all study groups.
Number of Participants Reporting Potential Immune-Mediated Diseases (pIMDs) | up to 14 months
  Number and percentage of patients reporting pIMDs from first vaccination up to study end for all study groups.
Number of Participants with Serious Adverse Events (SAEs) | up to 14 months
  Number and percentage of patients reporting SAEs and fatal SAEs from first vaccination up to study end for all study groups.
Number of Herpes Zoster Events | up to 14 months
  Number of cases of suspected HZ from study entry to last follow up date.
Number of Participants Reporting Complications from HZ | up to 14 months
  Number and percentage of patients reporting any complications of HZ reported as AEs from study entry to last follow up date.
Number of Participants reporting disease flares of IBD | baseline, Visit 1 (day 1), Follow-Up 2 (up to 29 days), Visit 2 (up to 90 days), Visit 3 (up to 140 days on study), Visit 4 (up to 360 days)
  Number and percentage of patients reporting disease flares of IBD in both study groups which will be assessed by monitoring disease activity using the Short Crohn's Activity Index (SCAI) for patients with Crohn's disease or the Simple Clinical Colitis Activity Index (SCCAI) questionnaire for patients with Ulcerative colitis at the baseline visit V1, Follow up 2 (FU2), V2, V3, and V4 visit.

OTHER OUTCOMES:
Number of gE-specific CD4 cells expressing at least 2 activation markers | Visit 1 (day 1), Visit 3 (up to 140 days on study), Visit 4 (up to 360 days)
  The number of gE-specific CD4 cells expressing at least 2 activation markers at V3 and at V4 compared to V1.
Vaccine response rate (VRR) in patients on JAKs | Visit 3 (up to 140 days on study)
  VRR with exact 95% CIs at V3.
Seropositivity rate in patients on JAKs | Visit 1 (day 1), Visit 3 (up to 140 days on study), Visit 4 (up to 360 days)
  Seropositivity rate with exact 95% CI at V1, V3, and V4
Geometric Mean Concentrations of Anti-gE Antibodies in Patients on JAKs | Visit 1 (day 1), Visit 3 (up to 140 days on study), Visit 4 (up to 360 days)
  Anti-gE antibody concentrations expressed as GMC with 95% CI at V1, V3, and V4 in patients on JAK's.
Geometric Mean Concentrations of Anti-gE Antibodies by Alpha Diversity of Microbiome | Visit 3 (up to 140 days on study)
  Anti-gE antibody concentrations expressed as GMC with 95% CI at V3 by alpha diversity of microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, MS, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Mayo Clinic, Jacksonville, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - New York University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - UW Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No